CLINICAL TRIAL: NCT05136573
Title: Quality Association
Brief Title: Exercises on CIPN, Fatigue, and Quality of Life in Colon Cancer Patients Receiving Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chi Mei Medical Hospital (Other)
Responsible Party: Principal Investigator, Chong-Chi Chiu, Center for quality management, Chi Mei Medical Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Chi Mei
Record Dates: First submitted 2021-11-02; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Experimental Study Designs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined Exercises on Symptoms of CIPN, Fatigue, and Quality of Life in Colon Cancer Patients (Experimental): The control group received routine care and maintenance of general daily activities; the experimental group received routine care and maintenance of general daily activities, and also received combined exercises
  Interventions: Behavioral: Combined Exercises

INTERVENTIONS:
Behavioral: Combined Exercises — Combined Exercises

SUMMARY:
Objective:

Cancer is one of the biggest global health threats. The incidence and mortality of colorectal cancer (CRC) are increasing. The treatment of CRC is mainly surgical resection, and the standard treatment of metastatic colorectal cancer is Oxaliplatin chemotherapy, which is mainly a platinum agent (Alkylating agent). Oxaliplatin can exert its anti-cancer therapeutic effect by binding to cell DNA, and become toxic to neurons, damaging large and small fibers outside the brain and spinal cord. Causes peripheral neuropathy, which seriously affects the quality of life of patients. The purpose to develop the interventional and investigate intervention by exercise program of CRC patients with regard to the improvement effect of peripheral neuropathy, fatigue and quality of life during the treatment.

Methods:

Experimental study designs were used, and samples were taken from a regional teaching hospital. The control group received routine care and maintenance of general daily activities; the experimental group received routine care and maintenance of general daily activities, and also received combined exercises, balance training and resistance exercises twice a week, 60 minutes each time, plus weekly 5 walking exercises, 30 minutes each time, for a total of 12 weeks, of which the exercise training during chemotherapy and hospitalization is performed under the supervision of the investigator, and 1 balance training and resistance exercise are performed for 60 minutes each time to ensure that the patient performs. The correctness and safety of exercises, and balance training and resistance exercises in combination with the home style. During the home exercises, the researchers will give weekly telephone interviews to understand the patient's exercise status, and indeed achieve the balance training and resistance exercises twice a week. All measurement tools and methods are implemented in accordance with consistent standard operations. The control group took pre-tests when the case was closed, without interventional measures, but also performed post-tests in the same way as the experimental group at 6 weeks, 8 weeks, 10 weeks, and 12 weeks in the interventional experimental group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with colon cancer, were getting chemotherapeutic drugs with oxaliplatin.

Exclusion Criteria:

* bone metastasis, lower extremity lymphedema, cognitive dysfunction, musculoskeletal problems,and diabetic.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
FACT/GOG | 12 weeks
  FACT/GOG-CIPN
EORTC QLQ-C30 | 12 weeks
  qulity of life

IPD SHARING:
Plan to Share IPD: No